CLINICAL TRIAL: NCT06217744
Title: Mental Health Literacy and Academic Performance - A Randomized Clinical Trial
Brief Title: Mental Health Literacy and Academic Performance
Acronym: MHLAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MHEALTHACAD
Record Dates: First submitted 2023-12-18; First posted 2024-01-22 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Wellness 1
Keywords: adolescents; randomized clinical trial; mental health; resilience; youth
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: cluster RCT, with students nested into classrooms (level of randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated Intervention (Experimental): The intervention will last for 3 months, with two psychoeducational modules delivered per month.
  Interventions: Behavioral: Automated Intervention
- Blended Intervention (Experimental): The intervention will last for 3 months, with two psychoeducational modules delivered per month. In addition, regular synchronous or asynchronous psychoeducational sessions conducted by a licensed psychologist will be held with the participants.
  Interventions: Behavioral: Blended Intervention
- Waitlist (No Intervention): This group will undergo the evaluations on the same schedule like the active groups. No intervention will be done.

INTERVENTIONS:
Behavioral: Automated Intervention — Participants will receive 6 psychoeducational modules design to increase mental health literacy: Module 1: The Stigma of Mental Illness, Module 2: Understanding Mental Health and Mental Illness, Module 3: Information on Specific Mental Illnesses, Module 4: Experiences of Mental Illness, Module 5: Seeking Help and Finding Support, Module 6: The Importance of Positive Mental Health.
  Arms: Automated Intervention
Behavioral: Blended Intervention — Participants will receive the same materials as the Automated Intervention, as well as the possibility to attend psychoeducational sessions held by licensed psychologists.
  Arms: Blended Intervention

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an intervention designed to promote mental health literacy in adolescents. The main questions it aims to answer are:

1. Whether this intervention can have an impact on mental health
2. Whether this intervention can have an impact on fostering academic performance, particularly in disadvantaged students (i.e., academic resilience)
3. Whether this intervention will have differential effectiveness as a function of the delivery format (psychoeducational materials only versus blended)

Participants will receive either an online, automated intervention consisting of psychoeducational materials delivered at predetermined intervals (automated), or the same but with the addition of synchronous or asynchronous psychoeducational sessions held by a licensed psychologist (i.e., blended).

These two conditions will also be compared to a Waitlist, to test if the interventions perform better than no treatment.

DETAILED DESCRIPTION:
A Randomized Clinical Trial was designed, involving comparisons at three time-points (pre-intervention, post-intervention, and follow-up) between: (a) Automated delivery of the intervention, (b) Blended format of the intervention, (c) Waitlist (matched control group). Participants will be randomly allocated to one of these three arms, with randomization done at the classroom level.

Appropriate methods for two-level-designs were used to determine sample size requirements for a cRCT with 4 cluster groups (i.e. classrooms) per experimental condition, 22 participants per cluster. For a linear mixed-effects model, a sample size of approximately 88 participants per experimental condition for a total sample size of 264 was sufficient to achieve 80% power to detect an effect size of Cohen's d = 0.4 at an alpha level of 0.05.

Mental health symptomatology (screening items, Attention Deficit/Hyperactivity Disorder (ADHD), depression, anxiety, social anxiety, Posttraumatic Stress Disorder (PTSD), eating disorders), adverse childhood experiences, bullying, social support, mental health stigma, help-seeking, social media engagement, digital addiction, and academic performance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in High School

Exclusion Criteria:

* Younger than 14 or older than 18

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Academic Performance - reading | up to 3 months
  Reading comprehension will be assessed with a standardized test for Romanian language, which were sourced from the pool of items from the Progress in International Reading Literacy Study (PIRLS). The test will consist of 26 items, with difficulties ranging from easy to difficult. Higher scores indicate greater academic performance.
Academic Performance - mathematics | up to 3 months
  Performance in mathematics will be assessed with a standardized test, sourced from the TIMSS, a platform specializing in standardized educational assessment in Romania. The test will consist of 26 items, with difficulties ranging from easy to difficult. Higher scores indicate greater academic performance.
Depressive symptomatology | up to 3 months
  The Patient Health Questionnaire-9 Depression Scale (PHQ-A, Johnson et al., 2002) is the adolescent-adapted version of the Patient Health Questionnaire and contains ten items. Scores range from 0 to 30 and a higher score is representative of a worse outcome.
Anxiety symptomatology | up to 3 months
  The Anxiety Rating scale (Spitzer et al., 2011) consists of eight items, with scores ranging from 0 to 24 and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Social anxiety symptomatology | up to 3 months
  The Severity Measure for Social Anxiety Disorder (SMSAD 11-17) is a ten-item instrument for children and adolescents (Carlton et al., 2022), with scores ranging from 0 to 50, with higher scores being indicative of a worse outcome.
Posttraumatic stress symptomatology | up to 3 months
  Posttraumatic Stress The Post Traumatic Symptom scale (Nedelcea et al., 2022) consists of 37 items. The first part of the scale presents a series of 17 stressful situations and participants are asked to indicate whether they have been exposed to one or more of these events in their lifetime. The last 20 items refer to the individual's reaction after experiencing a stressful situation. Scores range from 0 to 80, with higher scores indicating a worse outcome.
Eating Disorder symptomatology | up to 3 months
  The NEDA Eating Disorder Screening Tool (Fitzsimmons-Craft et al., 2019) is composed of 14 items. The first 11 items address different aspects of eating behavior and/or self-image. These contain multiple response options, with participants being guided to choose the one that suits them. The last three items refer to information about height, lowest weight in the last year and current weight. Higher scores indicate higher symptomatology.
Perceived social support | up to 3 months
  The Perceived Social Support Questionnaire (Kliem et al., 2015) contains six items, measured on a five-point Likert-type scale, where 1 = Does not fit me at all and 5 = Fits me extremely well. Scores range from 6 to 30, with higher scores indicative of a better outcome.

OTHER OUTCOMES:
Help seeking | up to 3 months
  The Attitudes Toward Seeking Professional Psychological Help - Short Form (Fischer & Farina, 1995) instrument assesses attitudes towards seeking specialized psychological help. It consists of ten items and participants are asked to express the extent to which they agree with the statements. Scores range from 0 to 30 and higher scores are indicative of a better outcome.
Mental health stigma | up to 3 months
  The Peer Mental Health Stigmatization Scale (McKeague et al., 2015) assesses stigmatizing attitudes of people experiencing mental health problems. It is composed of 24 items and participants are asked to express the extent to which they agree with the items. cores range from 0 to 96, with higher scores being indicative of a better outcome.
Bullying | up to 3 months
  Bullying will assessed with the six items used in the World Mental Health Initiative. The items refer to times when someone is intentionally hurt or scared by a peer in the school setting, on the internet and in close relationships. Scores range from 0 to 24, with higher scores indicative of a worse outcome.
Social media engagement | up to 3 months
  Social Media engagement will be measured with the Social Media Engagement Questionnaire (SMEQ; Przybylski et al., 2013). The questionnaire contains 5 items measured on an 8-point Likert scale (0 = not one day; 7 = every day). Higher scores represent higher engagement with social media. Scores range from 0 to 35, with higher scores indicative of a worse outcome.
Digital addiction | up to 3 months
  Digital Addiction will be measured with the Digital Addiction Scale for Teenagers (DAST; Seema et al., 2022). This is a 10-item instrument measured on a 7-point Likert scale ranging from never to very often. Scores range from 0 to 60, with higher scores indicative of a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — University of Bucharest
Locations (1):
- University of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giosan C, Pana A, Cosmoiu A, Chira AM, Toma AM, Papasteri CC, Nedelcea C, Popoviciu C. Mental health literacy and academic performance (MHLAP) in high school students: a randomized clinical trial protocol. Trials. 2024 Jun 27;25(1):419. doi: 10.1186/s13063-024-08270-y. PMID 38937769